CLINICAL TRIAL: NCT05866263
Title: Investigation of the Effect Of Green Walking and Intelligence Games on the Cognitive Skills of Individuals Between the Ages of 50-70 Survived COVID-19 Disease
Brief Title: Investigation of the Effect on Cognitive Skills of COVID-19 Survivors
Acronym: Cognitive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayburt University (Other)
Collaborators: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Zahide Akeren, Lecturer, Bayburt University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BayburtU; Karadeniz Technical University (Other: Karadeniz Technical University)
Record Dates: First submitted 2023-04-07; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
Keywords: COVID-19; Attention; Nature; Memory; Intelligence; Walking
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: COVID-19 on an outpatient basis were completed with 40 individuals, 20 of which were in the green walking and intelligence game group and 20 were in the control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- green walking and intelligence game group (Experimental): The randomized controlled study to examine the effects of green walking and intelligence games on the cognitive skills of individuals aged 50-70 years who had COVID-19 on an outpatient basis were completed with 40 individuals, 20 of which were in the green walking and intelligence game group
  Interventions: Other: green walking and intelligence gam
- control group (Active Comparator): The randomized controlled study to examine the effects of green walking and intelligence games on the cognitive skills of individuals aged 50-70 years who had COVID-19 on an outpatient basis were completed with 40 individuals, 20 of which were in the 20 were in the control group
  Interventions: Other: green walking and intelligence gam

INTERVENTIONS:
Other: green walking and intelligence gam — The randomized controlled study to examine the effects of green walking and intelligence games on the cognitive skills of individuals aged 50-70 years who had COVID-19 on an outpatient basis were completed with 40 individuals, 20 of which were in the green walking and intelligence game group and 20 were in the control group.
  Other Names: control

SUMMARY:
Investigation of the Effect Of Green Walking and Intelligence Games on the Cognitive Skills of Individuals Between the Ages of 50-70 Survived COVID-19 Disease

The randomized controlled study to examine the effects of green walking and intelligence games on the cognitive skills of individuals aged 50-70 years who had COVID-19 on an outpatient basis were completed with 40 individuals, 20 of which were in the green walking and intelligence game group and 20 were in the control group.

DETAILED DESCRIPTION:
The data were collected in Erzincan Tercan State Hospital between January-May 2022, "Patient Information Form," "Montreal Cognitive Assessment Implementation Guideline," "Brain Games (Brain Games-Memory Thinking and Brain Exercise) Information Leaflet," "Hiking Information Brochure," and "Experimental Group Follow-up Form" by the "Montreal Cognitive Assessment Scale" applied as a pre-test. As an initiative, the green walking and intelligence game group was given a 30-minute nature walk three days a week for a month and a 15-minute intelligence game practice every day. Then, the "Montreal Cognitive Assessment Scale" was applied as a post-test.

ELIGIBILITY:
Inclusion Criteria:

* Electronic records and contact information (address, telephone) of individuals who were diagnosed with COVID-19 in Erzincan Tercan State Hospital and whose COVID-19 test became negative within one year after being placed in home quarantine with outpatient treatment,
* Individuals are between the ages of 50-70,
* A score of 20 or less on the Montreal Cognitive Assessment Scale,
* To be at least primary school graduate,
* Being residing in the Tercan district of Erzincan,
* Being able to perform self-care activities independently,
* Good general condition,
* Having a smart phone or having a smart phone in one person in the household,
* For individuals in the trekking and intelligence game group, for one month It indicates that there is no harm in taking a nature walk for 30 minutes three days a week, having the approval of the physician.
* Agreeing to participate in the research.
* Exclusion Criteria for Research
* Positive COVID-19 (PCR) test result,
* Being visually and hearing impaired,
* Having a balance problem
* Using a cane or walker while walking,
* Being dependent on a bed or a wheelchair,
* Parkinson's, dementia, Alzheimer's diagnosis,
* Getting a diagnosis of cancer,
* Having a history of central nervous system disease that may cause cognitive dysfunction (stroke, head trauma, tumor, epilepsy, movement disorder diseases),
* Using antipsychotics, antidepressants, mood stabilizers, antiepileptics, benzodiazepines and medications that may interfere with the evaluation,
* Having undergone any surgery to prevent walking,
* Having a condition that prevents walking (musculoskeletal problems, joint problems, fracture, neuropathy, chronic severe pain, loss of limb).
* Exclusion Criteria
* Do not be hospitalized for any reason,
* Change of residence, emigration, death,
* Having an infection that requires isolation,
* Worsening of the general condition,
* Inclusion in another aerobic exercise program,
* Unwillingness to continue research.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Investigation on the Cognitive Skills of Individuals Between the Ages of 50-70 Survived COVID-19 Disease | for a month
  Examine the effects of green walking and intelligence games on the cognitive skills of individuals aged 50-70 years who had COVID-19 on an outpatient basis were completed with individuals

CONTACTS AND LOCATIONS:
Overall Officials: ZAHİDE AKEREN, Principal Investigator — Bayburt University
Locations (1):
- Erzincan Tercan State Hospital, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Application of the Experimental Group Follow-up Form The nature of the individuals in the green walking and intelligence game group were recorded by the researcher on the Experiment Group Follow-up Form 12 times, three days a week, on the day of the trek. In addition, the situation of playing the intelligence game of this group of individuals is a test for each individual. In addition, the state of playing intelligence games of this group of individuals was recorded by the researcher in the Experimental Group Follow-up Form by making 30 phone calls, including once a day for a month, for each individual.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: January-May 2022
Access Criteria: The work has been completed and is not accessible.

REFERENCES:
- [Result] Nouchi R, Taki Y, Takeuchi H, Hashizume H, Nozawa T, Kambara T, Sekiguchi A, Miyauchi CM, Kotozaki Y, Nouchi H, Kawashima R. Brain training game boosts executive functions, working memory and processing speed in the young adults: a randomized controlled trial. PLoS One. 2013;8(2):e55518. doi: 10.1371/journal.pone.0055518. Epub 2013 Feb 6. PMID 23405164
- See also: https://pubmed.ncbi.nlm.nih.gov/23405164/ — http://pubmed.ncbi.nlm.nih.gov/23405164/
- Available data/document: Informed Consent Form — https://pubmed.ncbi.nlm.nih.gov/23405164/
- Available data/document: Study Protocol — https://pubmed.ncbi.nlm.nih.gov/23405164/